CLINICAL TRIAL: NCT05445271
Title: The Effects of Endotracheal Intubation or Laryngeal Mask Applications on Optic Nerve
Brief Title: Optic Nerve Sheath Diameter in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Feyza Calisir, Assistant professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2018/01-28
Record Dates: First submitted 2022-06-29; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Optic Nerve Sheath Neoplasm; Intracranial Pressure Increase; Intubation Complication; Airway Complication of Anesthesia
MeSH Terms: conditions — Optic Nerve Neoplasms; Intracranial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): 30 patients who will be intubated with a video laryngoscope and who meet the inclusion criteria are randomly selected by lottery method. After obtaining the consent of the patient's family, the patient is taken to the operating room and monitored. 5 minutes after sedation with 1 mg midazolam, the optic nerve sheath diameter of both eyes is measured with a linear ultrasound probe and recorded (T0). 5 minutes after the patient is intubated with a video laryngoscope, the optic nerve sheath diameter of both eyes is measured and recorded (T1). After the patient's extubation at the end of the case, the optic nerve sheath diameter of both eyes is measured and recorded (T2). Vitals (pulse, blood pressure, saturation) involved in T0, T1 and T2 processes are recorded.
  Interventions: Diagnostic Test: Optic nerve sheath diameter measurement with linear ultrasound
- Group 2 (Active Comparator): 30 patients who will be intubated with a normal laryngoscope and who meet the inclusion criteria are randomly selected by lottery method. After obtaining the consent of the patient's family, the patient is taken to the operating room and monitored. 5 minutes after sedation with 1 mg midazolam, the optic nerve sheath diameter of both eyes is measured with a linear ultrasound probe and recorded (T0). 5 minutes after the patient is intubated with a normal laryngoscope, the optic nerve sheath diameter of both eyes is measured and recorded (T1). After the patient's extubation at the end of the case, the optic nerve sheath diameter of both eyes is measured and recorded (T2). Vitals (pulse, blood pressure, saturation) involved in T0, T1 and T2 processes are recorded.
  Interventions: Diagnostic Test: Optic nerve sheath diameter measurement with linear ultrasound
- Group 3 (Active Comparator): 30 patients who will be ventilated with a laryngeal mask airway (LMA) and who meet the inclusion criteria are randomly selected by lottery method. After obtaining the consent of the patient's family, the patient is taken to the operating room and monitored. 5 minutes after sedation with 1 mg midazolam, the optic nerve sheath diameter of both eyes is measured with a linear ultrasound probe and recorded (T0). The optic nerve sheath diameter of both eyes is measured and recorded 5 minutes after LMA is placed on the patient (T1). After the patient's extubation at the end of the case, the optic nerve sheath diameter of both eyes is measured and recorded (T2). Vitals (pulse, blood pressure, saturation) involved in T0, T1 and T2 processes are recorded.
  Interventions: Diagnostic Test: Optic nerve sheath diameter measurement with linear ultrasound

INTERVENTIONS:
Diagnostic Test: Optic nerve sheath diameter measurement with linear ultrasound — In this study, we aimed to show whether endotracheal intubation or LMA applications with optic nerve sheath diameter measurement, which is a completely non-invasive method, have effects on intracranial pressure.

SUMMARY:
Endotracheal intubation and laryngeal mask are generally applied to secure the airway during general anesthesia. There is a widespread opinion among anesthesiologists that endotracheal intubation increases intracranial pressure. Since there were no non-invasive methods measuring intracranial pressure in the past, adequate studies on this subject could not be done. With this measurement, we aimed to show whether ETT or LMA applications have effects on intracranial pressure.

DETAILED DESCRIPTION:
In normal pediatric patients with closed fontanelles, the contents of the central nervous system are almost compressed into the skull and spinal canal. Intracranial pressure is created and constant by the total volume of brain, CSF, and blood within the skull. Increased intracranial pressure can be measured with an intraventricular catheter, transducers, and a subarachnoid bolt. By measuring the diameter of the optic nerve sheath with ultrasonography, we can find out whether there is an increase in intracranial pressure non-invasively.

Endotracheal intubation and laryngeal mask are generally applied to secure the airway during general anesthesia. There is a widespread opinion among anesthesiologists that endotracheal intubation increases intracranial pressure. Since there were no non-invasive methods measuring intracranial pressure in the past, adequate studies on this subject could not be done. With this measurement, we aimed to show whether ETT or LMA applications have effects on intracranial pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 2-18 years
2. Patients undergoing general anesthesia
3. Patients who agreed to be included
4. ASA I-III

Exclusion Criteria:

1. Those with any eye pathology
2. Those with intracranial pathology

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter measurement at pediatric patients | 6 months
  to show whether endotracheal intubation or LMA applications with optic nerve sheath diameter measurement, which is a completely non-invasive method, have effects on intracranial pressure.

IPD SHARING:
Plan to Share IPD: Undecided